CLINICAL TRIAL: NCT05086731
Title: THRIVE Smart - Leveraging Mobile Health to Improve Oral Chemotherapy Adherence Among Women With Breast Cancer
Brief Title: Mobile Health to Improve Oral Chemotherapy Adherence Among Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: NRG Oncology (Other); National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Ilana Graetz, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00002985; NCI-2021-09125 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EU5395-21 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2021-10-19; First posted 2021-10-21 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Localized Breast Carcinoma; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Triple-Negative Breast Carcinoma; Metastatic Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (SMRxT smart pill bottle) (Experimental): Patients receive a SMRxT smart pill bottle, report symptoms weekly, and receive reminders for missing or incorrect dose for standard of care 3-week capecitabine/Xeloda treatment cycles.
  Interventions: Other: Informational Intervention; Other: Medical Device Usage and Evaluation; Other: Quality-of-Life Assessment; Other: Survey Administration
- Group II (standard of care) (Active Comparator): Patients receive a SMRxT smart pill bottle and standard of care.
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
  Arms: Group II (standard of care)
Other: Informational Intervention — Receive reminders
  Arms: Group I (SMRxT smart pill bottle)
Other: Medical Device Usage and Evaluation — Receive a SMRxT smart pill bottle
  Arms: Group I (SMRxT smart pill bottle)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates the feasibility and acceptability of a mobile health device in improving oral chemotherapy adherence in women with triple negative breast cancer that has not spread to other places in the body (non-metastatic). A mobile health device, called SMRxT smart pill bottle may help doctors to remind patients to take medicine on time and monitor their symptoms.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Feasibility. II. Acceptability. III. Capecitabine/Xeloda adherence.

EXPLORATORY OBJECTIVES:

I. Symptom burden. II. Patent physician communication. III. Quality of life. IV. Self-efficacy for managing symptoms.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive a SMRxT smart pill bottle, report symptoms weekly, and receive reminders for missing or incorrect dose for standard of care 3-week capecitabine/Xeloda treatment cycles.

GROUP II: Patients receive standard of care.

After completion of study, patients are followed up for 90 days after the initiation of capecitabine/Xeloda.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Breast cancer
* English speaking
* New or existing prescription for capecitabine/Xeloda
* Willingness and ability of the subject to comply with study procedures
* Have a mobile phone with text message
* Evidence of an online informed consent indicating that the subject is aware of the risk and benefits of study participation

Exclusion Criteria:

* Those who do not receive their capecitabine/Xeloda prescription until a month after enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status > 2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Medication adherence | From baseline up to 90 days
  Proportion of times each patient took her scheduled medication during the 3-month study. For each patient, will operationalize adherence as the number of times that the pill monitor recorded a dose taken for each day that the patient was in the study and supposed to take the pill. Days during which patients were off cycle, advised by their provider to temporarily stop the medication, or hospitalized will be deducted from the total days in the study.

SECONDARY OUTCOMES:
End-user engagement by patients and their oncology team | From baseline up to 90 days
  Will measure patient's use of the smart pill bottle, their response to weekly symptoms text message questions, response to the smart reminders, and response to the adherence reason text message question. In addition, will also measure and evaluate the provider response to any adherence or symptom alerts triggered during the intervention.
Acceptability | From baseline up to 90 days
  Will be measured using survey questions about the intervention after the 90-day intervention. Acceptability and usability will be determined using the System Usability Scale.

OTHER OUTCOMES:
Symptom burden | From baseline up to 90 days
  Will be measured using an adapted version of the National-Comprehensive Cancer Network Functional Assessment of Cancer Therapy Breast Cancer Symptom index (NCCN-FACT FBSI-16).
Self-efficacy for managing symptoms | From baseline up to 90 days
  Will be measured by 4-item PROMIS Item Bank version 1.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Graetz, PhD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (4):
- United States (4):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia

DOCUMENTS (1):
  • Informed Consent Form (2022-06-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT05086731/ICF_000.pdf